CLINICAL TRIAL: NCT00167869
Title: LACTOPRES:Study on the Effect of Dairy Peptides on Blood Pressure in Untreated Hypertensive Subjects.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: Unilever R&D (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: METC-WU 04/04
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure; dairy peptides; bioactive peptides; randomized controlled trial
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Behavioral: dairy peptides

SUMMARY:
Hypertension is an increasingly important medical and public health issue. Literature suggests that there may be a role for dairy foods in the prevention and treatment of hypertension. Recently, it has been suggested that several peptides in milk proteins could have blood pressure lowering properties. LACTOPRES is a randomised, double-blind parallel trial to assess the blood pressure effect of an increased intake of dairy peptides in humans.

ELIGIBILITY:
Inclusion Criteria:

* systolic blood pressure >= 140 mmHg
* BMI between 18 and 32 kg/m2
* apparently healthy

Exclusion Criteria:

* antihypertensive medication
* medically prescribed or slimming diet
* lactating, pregnant
* irregular pulse

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135
Dates: Start 2004-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Frans J Kok, PhD, Principal Investigator — Wageningen University - Division of Human Nutrition
Locations (1):
- Wageningen University, Division of Human Nutrition, Wageningen, Netherlands

REFERENCES:
- See also: Division of Human Nutrition, Wageningen University — http://www.humannutrition.nl